CLINICAL TRIAL: NCT06297330
Title: Determining the Influence of an Intervention Program Based on Sleep Improvement and Fatigue Reduction Among Medical Students.
Brief Title: Sleep for Optimal MEdical StudentS (PROMESS)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Research on Healthcare Performance Lab U1290 (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: PROMESS - SLEEP
Record Dates: First submitted 2024-02-29; First posted 2024-03-07 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-02

CONDITIONS: Health Behavior; Health-Related Behavior; Sleep; Sleep Disorder; Fatigue
Keywords: Health; Student; Curriculum; Behaviour; Medical; Sleep; Fatigue
MeSH Terms: conditions — Health Behavior; Sleep Wake Disorders; Fatigue; Behavior | interventions — Sleep

STUDY DESIGN:
Intervention Model Description: All volunteers will receive an intervention program based on sleep improvement and fatigue reduction.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sleep intervention (Experimental): One arm : All volunteers will receive a sleep management intervention.
  Interventions: Behavioral: Sleep

INTERVENTIONS:
Behavioral: Sleep — The sleep management intervention will consist of three individual sessions, each lasting one hour, with approximately 15 days between each session. The sessions will be scheduled as follow: week 5 and 6 (session 1), week 7 and 8 (session 2), week 9, 10, and 11 (session 3). During these sessions, subjective and objective indicators related to the sleep and fatigue levels will be recorded to assess the progress of each student.

SUMMARY:
Medical students have been shown to have a greater prevalence of poor sleep leading to poorer quality of life than other groups of students. Among medical students, poor sleep quality and insomnia have been associated with higher level of stress, as well as poorer academic performance. Our field surveys carried out in 2022 and 2023 at the Lyon Est medical school make the same alarming observation. They revealed that 53% of students had significant sleep problems.They also showed that students presented high levels of physical and mental fatigue. It is expected that these disorders will significantly degrade their quality of life as well as their health. Indeed, lack of sleep is associated with serious health problems such as illnesses cardiovascular or immune system deficiencies.

The PROMESS - SLEEP project aims to offer solutions to students to improve their sleep during their medical studies. It responds to a demand expressed by students: our field study showed that 40% of 4th year students declared being "very interested and/or interested" in following an intervention that aimed at improving sleep. An early knowledge of sleep optimization tools would allow students to quickly acquire the tools necessary to cope with the difficult conditions encountered during their training and lives of future doctors.The objective of this study is to determine the influence of an intervention program based on sleep improvement and fatigue reduction among medical students.

DETAILED DESCRIPTION:
Our project aims to help future healthcare professionals to adopt health-promoting behaviors during their studies in a preventive approach. This support will be provided through an intervention program based on sleep improvement and fatigue reduction during their curriculum. Specifically, 4th and 5th-year students at the Faculty of Medicine of Lyon Est will have the opportunity to participate in the PROMESS SLEEP project. This intervention will span 11 weeks. At the end of this period, we expect improvements in both subjective and objective indicators of sleep and fatigue.

METHODS.

PRE-INTERVENTION. Week 1-3. Students will undergo a two-hour session, during which, they will complete questionnaires on sleep and fatigue. Then, they will wear actimeters to monitor sleep during three weeks.

INTERVENTION. From week 5 to week 11. The intervention will consist of three individual sessions, each lasting one hour, with approximately 15 days between each session. Each session includes individual interview between a sleep expert and the participant (i.e.student).The sessions will be scheduled as follow: week 5 and 6 (session 1), week 7 and 8 (session 2), week 9, 10, and 11 (session 3). During the interview, the expert will realize an initial assessment of student sleep and fatigue levels and will give personalized goals to student. Subsequent sessions follow the same structure.

ELIGIBILITY:
Inclusion Criteria:

* Being a 4th-year or a 5th-year medical student at the Faculty of Medicine Lyon East during the academic year 2023-2024.
* Having read the information note.
* Having signed the written consent.

Exclusion Criteria: No exclusion criteria will be applied.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-11-11 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Perceived level of sleep troubles. Evolution of the score obtained at the Pittsburgh Sleep Questionnaire Inventory (PSQI). | From week 5 to week 11.
  The students level of sleep troubles will be assessed through the PSQI score ranging from 0 (none) to 21 (extreme). This score classified the presence or absence of sleep troubles. It can be divided into eight sub-scores (i.e., sleep quality, sleep latency, time spent in bed, sleep time, habitual sleep efficiency, sleep disturbance, use of sleeping medication and daytime dysfunction). The measure will be done every session, i.e. session 1 (week 5-6), session 2 (week 7-8) and session 3 (week 9,10,11).

SECONDARY OUTCOMES:
Perceived level of sleep troubles. Score obtained at the Pittsburgh Sleep Questionnaire Inventory (PSQI). | Week 1 (Pre-intervention)
  The students basal level of sleep troubles will be assessed through the PSQI questionnaire ranging from 0 (none) to 21 (extreme). One score is assessed and classified the presence or absence of sleep troubles. It can be divided into eight sub-scores (i.e quality, latence, time spent in bed, sleep time, sleep efficacy, daytime dysfunction, sleep troubles and pills). This measure will be done during the pre-interventional period at week 1.
Epworth Sleepiness scale. Score obtained at the Epworth Sleepiness scale. | Week 1 (Pre-intervention)
  The students basal level of diurnal sleepiness will be assessed through the Epworth Sleepiness scale ranging from 0 (none) to 24 (extreme). This measure will be done during the pre-interventional period at week 1.
Multidimensional Fatigue. Score obtained at the Multidimensional Fatigue Inventory (MFI). | Week 1 (Pre-intervention)
  The students basal level of fatigue will be assessed through the MFI questionnaire that covers various dimensions of fatigue, including general fatigue, physical fatigue, mental fatigue, reduced motivation, and reduced activity; ranging from 4 to 20. A total score can also be assessed (from 20 to 100). This measure will be done during the pre-interventional period at week 1.
Reduced composite scale of morningness. Score obtained at the reduced composite scale of morningness (RCSMS). | Week 1 (Pre-intervention)
  The students chronotype are assessed through the RCSMS. A total score can also be assessed (from 7 to 30). This measure will be done during the pre-interventional period at week 1.
Actimetry records. Time in Bed during the pre-intervention. | Week 1 (Pre-intervention)
  The objective students basal level of sleep will be accessed through the actimetry recordings.The time in bed (in hours/day) refers to the total duration between the time an individual gets into bed with the intention of sleeping and the time he/she get out of bed. It includes both the time spent asleep (total sleep time) and any periods of wakefulness while in bed. Essentially, it represents the total time allocated for sleep, regardless of whether the individual is actually sleeping during that time. This measure will be done during the pre-interventional period at week 1.
Actimetry records. Total sleep duration during the pre-intervention. | Week 1 (Pre-intervention)
  The objective students basal level of sleep will be accessed through the actimetry recordings. The total duration of sleep is obtained during a specified period, measured in hours/day. It represents the overall quantity of sleep obtained by an individual.This measure will be done during the pre-interventional period at week 1.
Actimetry records. Sleep efficiency during the pre-intervention. | Week 1 (Pre-intervention)
  The objective students basal level of sleep will be accessed through the actimetry recordings.The sleep efficiency is the ratio of total sleep time to the total time spent in bed, expressed as a percentage. It reflects how effectively one is sleeping during the time allotted for sleep. This measure will be done during the pre-interventional period at week 1.
Actimetry records. Sleep Onset Latency during the pre-intervention. | Week 1 (Pre-intervention)
  The objective students basal level of sleep will be accessed through the actimetry recordings. The sleep onset latency is the amount of time it takes for an individual to fall asleep after getting into bed, measured from the time the lights are turned off until sleep onset, reported in minutes.This measure will be done during the pre-interventional period at week 1.
Actimetry records. Wake after Sleep Onset during the pre-intervention. | Week 1 (Pre-intervention)
  The objective students basal level of sleep will be accessed through the actimetry recordings.The wake after sleep onset measures the total amount of time spent awake after initially falling asleep, reported in minutes. It reflects the disruptions in sleep continuity. This measure will be done during the pre-interventional period at week 1.
Actimetry records. Number of Awakenings during the pre-intervention. | Week 1 (Pre-intervention)
  The objective students basal level of sleep will be accessed through the actimetry recordings.The number of awakenings represents the frequency of brief awakenings during the sleep period. Each awakening may disrupt the continuity of sleep and impact sleep quality. This measure will be done during the pre-interventional period at week 1.
Actimetry records. Bedtime during the pre-intervention. | Week 1 (Pre-intervention)
  The objective students basal level of sleep will be accessed through the actimetry recordings. The bedtime is the time at which an individual goes to bed with the intention of sleeping. This measure will be done during the pre-interventional period at week 1.
Actimetry records. Mid-sleep point during the pre-intervention. | Week 1 (Pre-intervention)
  The objective students basal level of sleep will be accessed through the actimetry recordings.The mid-sleep point refers to the midpoint of an individual's sleep period. It is calculated by finding the halfway point between the time of sleep onset (when the individual falls asleep) and the time of sleep offset (when the individual wakes up). This measure will be done during the pre-interventional period at week 1.
Actimetry records. Sleep Onset time during the pre-intervention. | Week 1 (Pre-intervention)
  The objective students basal level of sleep will be accessed through the actimetry recordings.The sleep onset time refers to the time at which an individual falls asleep after initially getting into bed with the intention of sleeping, measured in minutes.This measure will be done during the pre-interventional period at week 1.
Actimetry records. Sleep Inertia during the pre-intervention. | Week 1 (Pre-intervention)
  The objective students basal level of sleep will be accessed through the actimetry recordings. The sleep inertia refers to the periods between wake-up time and get-up time, measured in minutes. This measure will be done during the pre-interventional period at week 1.
Actimetry records. Wake-up time during the pre-intervention. | Week 1 (Pre-intervention)
  The objective students basal level of sleep will be accessed through the actimetry recordings. The wake-up time refers to the time at which an individual awakens from sleep in the morning.This measure will be done during the pre-interventional period at week 1.
Actimetry records. Sleep regularity index during the pre-intervention. | Week 1 (Pre-intervention)
  The objective students basal level of sleep will be accessed through the actimetry recordings.The sleep regularity index is a measure that evaluates the consistency of an individual's sleep habits over a given period. It takes into account the regularity of bedtime and wake-up times on a daily basis. The higher the sleep regularity index, the more consistent and regular the individual's sleep habits are considered to be. This measure will be done during the pre-interventional period at week 1.
Multidimensional Fatigue. Evolution of the score obtained at the Multidimensional Fatigue Inventory (MFI) during the intervention. | From week 5 to week 11.
  The level of fatigue will be assessed through the MFI questionnaire that covers various dimensions of fatigue, including general fatigue, physical fatigue, mental fatigue, reduced motivation, and reduced activity; ranging from 4 to 20. A total score can also be assessed (from 20 to 100). The measure will be done every session, i.e. session 1 (week 5-6), session 2 (week 7-8) and session 3 (week 9,10,11).
Actimetry records. Evolution in Time in Bed during the intervention. | From week 5 to week 11.
  The measure will be done between every session, i.e. between session 1 (week 5-6) and session 2 (week 7-8) and between session 2 and session 3 (week 9,10,11).
Actimetry records. Evolution in Total sleep duration during the intervention. | From week 5 to week 11.
  The measure will be done between every session, i.e. between session 1 (week 5-6) and session 2 (week 7-8) and between session 2 and session 3 (week 9,10,11).
Actimetry records. Evolution in Sleep efficiency during the intervention. | From week 5 to week 11.
  The measure will be done between every session, i.e. between session 1 (week 5-6) and session 2 (week 7-8) and between session 2 and session 3 (week 9,10,11).
Actimetry records. Evolution in Sleep Onset Latency during the intervention. | From week 5 to week 11.
  The measure will be done between every session, i.e. between session 1 (week 5-6) and session 2 (week 7-8) and between session 2 and session 3 (week 9,10,11).
Actimetry records. Evolution in Wake after Sleep Onset during the intervention. | From week 5 to week 11.
  The measure will be done between every session, i.e. between session 1 (week 5-6) and session 2 (week 7-8) and between session 2 and session 3 (week 9,10,11).
Actimetry records. Evolution in Number of Awakenings during the intervention. | From week 5 to week 11.
  The measure will be done between every session, i.e. between session 1 (week 5-6) and session 2 (week 7-8) and between session 2 and session 3 (week 9,10,11).
Actimetry records. Evolution in Mid-sleep point during the intervention. | From week 5 to week 11.
  The measure will be done between every session, i.e. between session 1 (week 5-6) and session 2 (week 7-8) and between session 2 and session 3 (week 9,10,11).
Actimetry records. Evolution in Bed time during the intervention. | From week 5 to week 11.
  The measure will be done between every session, i.e. between session 1 (week 5-6) and session 2 (week 7-8) and between session 2 and session 3 (week 9,10,11).
Actimetry records. Evolution in Sleep Onset Time during the intervention. | From week 5 to week 11.
  The measure will be done between every session, i.e. between session 1 (week 5-6) and session 2 (week 7-8) and between session 2 and session 3 (week 9,10,11).
Actimetry records. Evolution in Sleep Inertia during the intervention. | From week 5 to week 11.
  The measure will be done between every session, i.e. between session 1 (week 5-6) and session 2 (week 7-8) and between session 2 and session 3 (week 9,10,11).
Actimetry records. Evolution in Wake-up Time during the intervention. | From week 5 to week 11.
  The measure will be done between every session, i.e. between session 1 (week 5-6) and session 2 (week 7-8) and between session 2 and session 3 (week 9,10,11).
Actimetry records. Evolution in Sleep regularity index during the intervention. | From week 5 to week 11.
  The measure will be done every session, i.e. session 1 (week 5-6), session 2 (week 7-8) and session 3 (week 9,10,11).
VAS - sleep quantity: Evolution of the score obtained at the 100-mm Visual Analogue Scale (VAS) assessing the quantity of sleep. | From week 5 to week 11.
  The students level of sleep quantity will be assessed on a 100-mm Visual Analogue Scale (VAS: "Over the past two weeks, how would you characterize your sleep?") ranging from 0 (quantity of sleep largely insufficient) to 100 (quantity of sleep largely sufficient). The measure will be done every session, i.e. session 1 (week 5-6), session 2 (week 7-8) and session 3 (week 9,10,11).
VAS - sleep quality. Evolution of the score obtained at the 100-mm Visual Analogue Scale (VAS) characterizing the sleep quality. | From week 5 to week 11.
  The students sleep quality will be assessed on a 100-mm Visual Analogue Scale (VAS: "Over the past two weeks, how would you characterize your sleep?") ranging from 0 (the worst quality of sleep possible) to 100 (the best quality of sleep possible). The measure will be done every session, i.e. session 1 (week 5-6), session 2 (week 7-8) and session 3 (week 9,10,11).
VAS - sleep fatigue. Evolution of the score obtained at the 100-mm Visual Analogue Scale (VAS) assessing the perceived level of fatigue. | From week 5 to week 11.
  The students level of fatigue will be assessed on a 100-mm Visual Analogue Scale (VAS: "Over the past two weeks, how would you characterize your physical and mental fatigue levels?") ranging from 0 (extreme fatigue) to 100 (absence total of fatigue).The measure will be done every session, i.e. session 1 (week 5-6), session 2 (week 7-8) and session 3 (week 9,10,11).
Advices given by the expert. Score obtained on a Likert scale ranging from 1 to 5 characterizing the nature of the advices given by the expert. | From week 5 to week 11.
  Following each session, the expert reported if he/she has given during the interview a specific advice according to apre-established list. For each pre-established advice, he/she has to report if :
  1. He/she didn't mention this
  2. He/she mentioned this but didn't directly advise it
  3. He/she mentioned this and recommended it
  4. He/she had set this in the goals
  5. The student was already doing it (positive reinforcement). The measure will be done every session, i.e. session 1 (week 5-6), session 2 (week 7-8) and session 3 (week 9,10,11).
Likert - expert estimation of student's achievements. Score obtained on a Likert scale ranging from 1 to 3 accessing if the expert estimates that the student has achieve the goals previously set. | From week 7 to week 11.
  The expert evaluates, from 0 to 3 (i.e. 0 : not achieved at all, 1: slightly achieved, 2: fairly well achieved, 3: well achieved) if he/she estimates that the student has achieve the goals previously set. The measure will be done at session 2 (week 7-8) and session 3 (week 9,10,11).
Likert - expert satisfaction. Scores obtained on a Likert scale ranging from 1 to 5 accessing the expert's satisfaction of his/her intervention. | From week 5 to week 11.
  The perceived level of the expert satisfaction ("Are you satisfied with the session you just realized?") will be accessed on a likert scale ranging from 1 (not at all satisfied) to 5 (very satisfied). The measure will be done every session, i.e. session 1 (week 5-6), session 2 (week 7-8) and session 3 (week 9,10,11).
Likert - expert level of comfort. Score assessing the expert comfort levels in participant relationships on a likert scale ranging from 1 to 5. | From week 5 to week 11.
  The perceived level of expert comfort of the relationship with the student ("How comfortable did you feel with the student?") will be accessed on a likert scale ranging from 1 (not at all comfortable) to 5 (very comfortable). The measure will be done every session, i.e. session 1 (week 5-6), session 2 (week 7-8) and session 3 (week 9,10,11).
Likert - expert estimation of the overall student's achievements. Score obtained on a Likert scale ranging from 1 to 5 accessing the expert's level of satisfaction on the student's progress. | Week 9-10-11
  The level of expert satisfaction of the student's progress ("Are you satisfied with the student's progress during the all intervention?") will be accessed on a likert scale ranging from 1 (not at all satisfied) to 5 (very satisfied). This measure will be done at the session 3, i.e. approximately at week 9,11,10.
Composite score - Student's satisfaction. Score ranging from 0 to 100 accessing the student's level of satisfaction of the all intervention. | Week 9-10-11
  The composite score will be the mean of two sub-scores :
  1. An intervention specific score. Mean of the scores obtained at the two 100-mm Visual Analogue Scales ranging from 0 (absolutely not) to 100 (completely) :
     * VAS: "Do you think the module has helped you to improve your sleep?"
     * VAS: "Do you think the module has helped you to decrease your fatigue?"
  2. An intervention general score. Mean of the scores obtained at the two 100-mm Visual Analogue Scales ranging from 0 (absolutely not) to 100 (completely) :
     * VAS :"Do you think the proposed goals were suitable for your daily life?"
     * VAS: "Do you think you can sustain the habit changes?" Theses measures will be done at the session 3, i.e. approximately at week 9,11,10.

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Schlatter, Dr., Principal Investigator — RESHAPE U1290 INSERM UCBL-LYON 1 Rockfeller, Lyon France.
Locations (1):
- RESHAPE, Lyon, France

REFERENCES:
- [Derived] Ruet A, Ndiki Mayi EF, Metais A, Valero B, Henry A, Duclos A, Lilot M, Rode G, Schlatter S. Determining the influence of a sleep improvement intervention on medical students' sleep and fatigue: protocol of the PROMESS-Sleep clinical trial. BMC Med Educ. 2025 Feb 19;25(1):267. doi: 10.1186/s12909-024-06422-x. PMID 39972313